CLINICAL TRIAL: NCT03840954
Title: Effects of Neuromuscular Electrical Stimulation in Muscle Architecture and Functionality of Patients After Acute Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20180460
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Stroke, Acute; Neuromuscular Electrical Stimulation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular Electrical Stimulation (Experimental): The experimental group will receive the application of NMES associated with conventional physiotherapy. After the NMES application, conventional physiotherapy will be performed. The exercises performed will be according to the patient's physical condition, and the conducts will always be performed seeking the maximum possible functional performance for the patient. The conducts adopted according to the standard routine of the HCPA stroke unit are: passive, active, assisted and / or active exercises; muscle stretching; selective hip extension; trunk stabilization training in sedestation; orthostasis training and walking training.
  Interventions: Other: Neuromuscular Electrical Stimulation
- Group Control (No Intervention): The control group will only receive conventional physiotherapy, composed of the same exercises performed in the experimental group.

INTERVENTIONS:
Other: Neuromuscular Electrical Stimulation — The application of NMES will be performed with the patient positioned in the supine position in the bed. Self-adhesive electrodes will be positioned at the motor points of the quadriceps and anterior tibial muscles respectively. A symmetrical biphasic pulsed current with a frequency of 80 Hz, a pulse width of 500 μs and an intensity at the motor threshold will be applied up to the maximum tolerated by the patient. ON and OFF time and total session time will be used according to protocol with progressive increase of the total intervention time and reduction of OFF time of the NMES. The device used will be the Neurodyn II model, manufactured by IBRAMED.
  Patients will receive NMES for as long as they remain hospitalized or for up to 3 weeks.
  Arms: Neuromuscular Electrical Stimulation

SUMMARY:
Introduction: Stroke is a sudden illness, responsible for important neurological and cognitive sequelae that can result in functional limitations and dependence. It is the leading cause of neurological impairment in young adults and resting-related muscle loss is one of the major factors involved. Early rehabilitation is essential for these patients and neuromuscular electrical stimulation (NMES) has been identified as an intervention alternative due to its known effects on the prevention of muscle loss in patients with various pathologies. Objective: To evaluate the effects of NMES associated with conventional physiotherapy compared to conventional physiotherapy on muscle thickness and functionality of patients with acute stroke. Methodology: This is a randomized clinical trial, which will be performed at the Emergency and Unit Unit of the Stroke of the Hospital de Clínicas of Porto Alegre (HCPA). Patients with acute stroke, with up to 72 hours of hospital admission, who present with lower limb force deficit due to the current stroke will be included. Patients will be randomized into two groups: intervention group, who will receive the application of NMES associated with conventional physiotherapy and control group, who will receive the conventional physiotherapy of the HCPA. NMES training will be applied once a day (30 minutes of application per session with an increase of five minutes each week and gradual reduction in OFF time), five days a week until hospital discharge or up to a maximum of three weeks. The following outcomes will be assessed before and after the intervention: quadriceps and tibial thickness and quality of the quadriceps and tibialis anterior, muscle strength, stroke severity, gait, functionality and disability.

DETAILED DESCRIPTION:
Stroke is the leading cause of neurological impairment in young adults, and early rehabilitation is essential for the recovery of these patients.

It is already known that muscle loss is one of the main factors responsible for functional disability and dependence in stroke survivors, being observed already in the acute phase and mainly in the lower limbs. The physiological mechanisms involved in stroke-related muscle loss, such as muscle inactivity, denervation, malnutrition, inflammation and metabolic disorders, among others have been reported in studies, but there is no consistent evidence regarding effective therapies to avoid muscle loss.

The NMES is already widely used for the prevention of muscular loss in patients with various pathologies. Studies have also reported the efficacy of NMES in patients with subacute or chronic stroke. In patients with acute stroke, the literature is rather scarce. The investigators are aware of only one study that evaluated the effects of NMES on muscle mass loss, but the authors did not evaluate the effects of this intervention on the physical performance or functionality of the patients. Thus, the investigators consider the importance of further studies to know the effects of NMES on muscle loss in patients with acute stroke and the need to evaluate the effects of NMES on the physical performance functionality of these patients aiming at the possibility of offering an intervention option precocious and effective for this population.

The objective of this study is to evaluate the effects of NMES associated with conventional physiotherapy compared to conventional physiotherapy in the muscular architecture and functionality of patients with acute stroke.

This is a randomized clinical trial in which the participants will be randomly divided into experimental group (EG) and control group (CG), being evaluated before and after the intervention.

The sample will be composed of hospitalized patients diagnosed with acute stroke at the Hospital de Clínicas de Porto Alegre (HCPA).

The estimated sample is 70 patients (35 in each group). Waiting for a 0.5 cm difference in muscle thickness between groups and a standard deviation of 0.68 and 2 of 0.80, with a significance level of 5%, 80% power.

Randomization will be performed through data generated by a computer program that presents the coded distribution. The sequence generation of the numbers to be randomized will be performed by a researcher blind to the study - after selection of the patients according to the eligibility criteria - keeping it confidential until the beginning of the intervention.

Data collect:

Socio-demographic data will be collected such as: age and sex; anthropometric variables: weight, height and BMI; and clinical data: stroke region, side of hemiparesis, comorbidities, complications during the hospitalization period (eg pneumonia, need for decompressive craniectomy), functional condition prior to the current stroke, time to start physical therapy, time to onset of NMES, total time of NMES, time to reach orthostasis and time to start ambulation. These data will be obtained through the review of medical records and interviews with patients or relatives.

Assessments: The evaluations described below will be performed within 72 hours of hospital admission and repeated at hospital discharge or within 21 days.

Assessment of muscle architecture - The assessment of muscle thickness will be performed in the femoral and tibial quadriceps muscles (TA). The images will be obtained by ultrasound using the Portable Ultrasound System (Vivid i®, GE) with a linear arrangement probe (60mm, 7.5 MHz - Vivid i®, GE). The same researcher (who will be blinded for the interventions) will do all the evaluations, which will be performed with the musculature at rest.

Muscle Strength Assessment: Manual Dynamometry, Medical Research Council (MRC)

Functional and Inability Assessment: Barthel's Index Modified

Walking assessment and functional capacity: Functional Ambulation Category (FAC)

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ischemic or hemorrhagic stroke performed by a neurologist based on clinical and neuroimaging characteristics;
* To present motor sequelae in the lower limb due to stroke.

Exclusion Criteria:

* Previous motor deficits
* Complete recovery of motor deficits before the initial evaluation;
* Conditions that prevent neuromuscular electrical stimulation such as skin lesions at the site of electrode placement, pacemaker and therapy intolerance.
* Time greater than 72 hours since hospitalization.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-08-30 (Estimated); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Quadriceps muscle thickness | three weeks
  Evaluated by muscular echography (cm)
Thickness of the anterior tibial muscle | three weeks
  Evaluated by muscular echography (cm)

SECONDARY OUTCOMES:
Functionality - Barthel Index for Activities of Daily Living | three weeks
  The score ranges from 0 to 100 points (90 to 100 - independent, 60 to 89 - slightly dependent, 40 to 59 - moderately dependent, 20 to 39 - severely dependent and less than 20 - totally dependent).
Muscle strength - Medical Research Council (MRC) Scale | three weeks
  The MRC score is obtained by evaluating 12 muscle groups in the upper extremities (wrist extensors, elbow flexors and abductors of the shoulder) and lower extremities (dorsal ankle flexors, knee extensors, and hip flexors). For each muscle group will be assigned a score between 0 (complete paralysis) and 5 (normal force), and the total score can vary between 0 up to 60 points.
Functional walking - Functional Ambulation Categories | three weeks
  Evaluates the degree of assistance required for ambulation. It distinguishes six categories for ambulation ability (1 to 3 - need for physical assistance during walking, 4 - requires only supervision and 5 and 6 - independent walking).
Dynamometry - Knee extension | three weeks
  Dynamometry (kg)
Dynamometry - ankle dorsiflexion | three weeks
  Dynamometry (kg)
Sit and stand up to 30 seconds | three weeks
  Assess the maximum number of times it is possible to get up and sit down in 30 seconds
Modified Rankin Scale | three weeks
  Evaluates the degree of disability and dependence in daily life with a score of 0: without any symptom at 6: death
10-meter walking test | three weeks
  Evaluates gait speed and cadence

CONTACTS AND LOCATIONS:
Overall Officials: Graciele Sbruzzi, doctor, Study Director — Federal University of Rio Grande do Sul
Locations (1):
- HCPA, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No